CLINICAL TRIAL: NCT05070897
Title: Health Literacy and Digital Health in Cancer Patients.
Acronym: LICAPA
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB 2021-04; 2021-A01725-36 (Other: ID-RCB number ANSM)
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: Health literacy; Digital health
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population A: 65 years old and more
  Interventions: Other: Questionnaires
- Population B: 18 to 64 years old
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — * Approved French version of the FCCHL scale
  * Questionnaire on the use of digital tools adapted from the questionnaire on digital tools

SUMMARY:
This is a multicentric, prospective, observational, transversal study, aiming to evaluate the health literacy of cancer patients using the approved French version of the Functional, Communicative and Critical Health Literacy (FCCHL) scale in 2 populations:

* Population A: patients age 65 and over treated in an oncology or oncogeriatric outpatient clinic, or seen in an oncology or oncogeriatric consultation.
* Population B: young patients age 18 to 64 treated in an oncology or outpatient clinic, or seen in an oncology consultation.

The following questionnaires:

* Approved French version of the FCCHL scale
* Questionnaire on the use of digital tools adapted from the questionnaire on digital tools,

will be completed once only. It will be completed by the participant during the oncology or oncogeriatric consultation or outpatient clinic appointment, in self-questionnaire mode or face to face, assisted if necessary by a family member or member of the medical team.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman.
2. Age ≥ 18 years.
3. Patient treated for cancer.
4. Patient who can read and understand French.
5. Patient seen in an oncology or oncogeriatric consultation or treated in an outpatient clinic.
6. Patient in treatment or about to start treatment that has been offered to them, from the announcement consultation to 2 years after the start of treatment

Exclusion Criteria:

1. Patient hospitalised for longer than 24 hours.
2. Patient with know cognitive impairment preventing them from answering the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in an oncology, or oncogeriatric consultation or treated in an oncology or geriatric outpatient clinic (not including full hospitalisation lasting ≥ 24h).
Sampling Method: Probability Sample
Enrollment: 1518 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pr Elene Paillaud, Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Population A: 65 years old and more ...
  Questionnaires: • Approved French version of the FCCHL scale
  • Questionnaire on the use of digital tools adapted from the questionnaire on digital tools
- Population B: 18 to 64 years old ... Questionnaires: • Approved French version of the FCCHL scale
  • Questionnaire on the use of digital tools adapted from the questionnaire on digital tools
Period: Overall Study
Arm/Group | Population A | Population B
Started | 781 | 737
Completed | 658 | 669
Not Completed | 123 | 68
Not completed — Protocol Violation | 123 | 68

BASELINE CHARACTERISTICS:
Groups:
- Population A: 65 years old and more
  Questionnaires: • Approved French version of the FCCHL scale
  • Questionnaire on the use of digital tools adapted from the questionnaire on digital tools
- Population B: 18 to 64 years old
  Questionnaires: • Approved French version of the FCCHL scale
  • Questionnaire on the use of digital tools adapted from the questionnaire on digital tools
- Total: Total of all reporting groups
Arm/Group | Population A | Population B | Total
Number analyzed (Participants) | 781 | 737 | 1518
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 737 | 737
  >=65 years | 781 | 0 | 781
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 74.9 [70 to 80] | 51.9 [46.0 to 60.0] | 63.7 [54.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 407 | 488 | 895
  Male | 374 | 249 | 623
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 781 | 737 | 1518
Living place [Count of Participants; unit: Participants]
  Home | 763 | 721 | 1484
  Nursing home | 6 | 3 | 9
  Other | 7 | 6 | 13
  Missing | 5 | 7 | 12
Do you live alone? [Count of Participants; unit: Participants]
  Yes | 243 | 159 | 402
  No | 531 | 565 | 1096
  Missing | 7 | 13 | 20
Area of residence [Count of Participants; unit: Participants]
  Urban | 439 | 385 | 824
  Rural | 287 | 288 | 575
  Missing | 55 | 64 | 119
Help for daily activites (neighbour, family, friends, medical professional) [Count of Participants; unit: Participants]
  Yes | 465 | 479 | 944
  No | 246 | 206 | 452
  Missing | 70 | 52 | 122
Cancer status [Count of Participants; unit: Participants]
  Localised | 233 | 286 | 519
  Advanced and/or metastatic | 547 | 448 | 995
  Not documented | 1 | 2 | 3
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Overall Score of ≤ 4 on the FCCHL Scale.
Description: Health literacy of cancer patients using the approved French version of the Functional, Communicative and Critical Health Literacy (FCCHL) scale. The FCCHL questionnaire includes 14 items, divided into 3 sub-scales, reflecting 3 health literacy skills (functional literacy, interactive literacy and critical literacy). The overall score will be calculated by determining the mean score for the 3 sub-scales. A score of ≤ 4 on the FCCHL scale, corresponds to a low level of health literacy. Each item of the FCCHL takes a score of 1 to 5 points. For each patient, a literacy score per sub-scale will be determined by calculating the number of points divided by the number of items on the sub-scale. The score can range from 1 to 5. The overall literacy score will be calculated as the mean of the 3 sub-scales. This score can range from 1 to 5.
  For functional scale, higher value represent worse outcome and for the other scale, a higher value represent a better outcome.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Population A | Population B
Number analyzed (Participants) | 658 | 669
Participants | 518 | 468

2. Secondary Outcome: Number et Percentage of Participants by Items of the Questionnaire on the Use of Digital Tools.
Description: The questionnaire on the use of digital tools will be described per item:
  * This questionnaire includes 10 items.
  * A Likert-type scale with five modalities of response is proposed (never, rarely, sometimes, often, always).
  * No overall score will be calculated.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Population A | Population B
Number analyzed (Participants) | 781 | 737
Participants
  Use of internet: Never | 232 | 39
  Use of internet: Rarely | 26 | 17
  Use of internet: Sometimes | 64 | 43
  Use of internet: Often | 156 | 133
  Use of internet: Always | 284 | 493
  Use of internet: Not available | 19 | 12
  Use of internet for you health: Never | 321 | 100
  Use of internet for you health: Rarely | 67 | 62
  Use of internet for you health: Sometimes | 152 | 179
  Use of internet for you health: Often | 128 | 231
  Use of internet for you health: Always | 86 | 149
  Use of internet for you health: Not available | 27 | 16
  Communication by email in daily life: Never | 278 | 76
  Communication by email in daily life: Rarely | 35 | 36
  Communication by email in daily life: Sometimes | 81 | 88
  Communication by email in daily life: Often | 154 | 203
  Communication by email in daily life: Always | 215 | 323
  Communication by email in daily life: Not available | 18 | 11
  Use a smartphone (with internet connection and applications): Never | 146 | 36
  Use a smartphone (with internet connection and applications): Rarely | 21 | 6
  Use a smartphone (with internet connection and applications): Sometimes | 45 | 13
  Use a smartphone (with internet connection and applications): Often | 91 | 62
  Use a smartphone (with internet connection and applications): Always | 460 | 612
  Use a smartphone (with internet connection and applications): Not available | 18 | 8
  Communication by texts in daily life: Never | 199 | 29
  Communication by texts in daily life: Rarely | 35 | 10
  Communication by texts in daily life: Sometimes | 70 | 40
  Communication by texts in daily life: Often | 147 | 139
  Communication by texts in daily life: Always | 316 | 510
  Communication by texts in daily life: Not available | 14 | 9
  Use a touch pad in daily life: Never | 454 | 265
  Use a touch pad in daily life: Rarely | 34 | 59
  Use a touch pad in daily life: Sometimes | 46 | 81
  Use a touch pad in daily life: Often | 62 | 94
  Use a touch pad in daily life: Always | 167 | 223
  Use a touch pad in daily life: Not available | 18 | 15
  Use a computer in daily life: Never | 274 | 78
  Use a computer in daily life: Rarely | 34 | 35
  Use a computer in daily life: Sometimes | 56 | 77
  Use a computer in daily life: Often | 110 | 165
  Use a computer in daily life: Always | 292 | 368
  Use a computer in daily life: Not available | 15 | 14
  Use a medical apps (on pad or smartphone): Never | 593 | 367
  Use a medical apps (on pad or smartphone): Rarely | 56 | 103
  Use a medical apps (on pad or smartphone): Sometimes | 69 | 113
  Use a medical apps (on pad or smartphone): Often | 26 | 87
  Use a medical apps (on pad or smartphone): Always | 22 | 55
  Use a medical apps (on pad or smartphone): Not available | 15 | 12
  Use connected objects (e.g. connected swatch, pedometer, etc.): Never | 650 | 512
  Use connected objects (e.g. connected swatch, pedometer, etc.): Rarely | 29 | 46
  Use connected objects (e.g. connected swatch, pedometer, etc.): Sometimes | 21 | 58
  Use connected objects (e.g. connected swatch, pedometer, etc.): Often | 33 | 55
  Use connected objects (e.g. connected swatch, pedometer, etc.): Always | 34 | 60
  Use connected objects (e.g. connected swatch, pedometer, etc.): Not available | 14 | 6
  Use online consultations or telemedicine: Never | 647 | 472
  Use online consultations or telemedicine: Rarely | 54 | 87
  Use online consultations or telemedicine: Sometimes | 50 | 120
  Use online consultations or telemedicine: Often | 6 | 29
  Use online consultations or telemedicine: Always | 12 | 20
  Use online consultations or telemedicine: Not available | 12 | 9
  Change yours habits and use online consultations or telemedicine since the beginning of COVID-19?: Never | 642 | 469
  Change yours habits and use online consultations or telemedicine since the beginning of COVID-19?: Rarely | 61 | 91
  Change yours habits and use online consultations or telemedicine since the beginning of COVID-19?: Sometimes | 36 | 105
  Change yours habits and use online consultations or telemedicine since the beginning of COVID-19?: Often | 18 | 42
  Change yours habits and use online consultations or telemedicine since the beginning of COVID-19?: Always | 13 | 23
  Change yours habits and use online consultations or telemedicine since the beginning of COVID-19?: Not available | 11 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study
Description: Adverse events were not collected for this study
Arm/Group | Population A | Population B
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT05070897/Prot_001.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT05070897/SAP_002.pdf